CLINICAL TRIAL: NCT06563180
Title: Impact of Climate Changes on Women's Health in Al Dakahlya Governorate, Egypt
Acronym: Women
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Basma Wageah Mohamed Mohamed Elrefay, Lecturer of obstetrics and gynaecology Nursing, Faculty of nursing- Delta University for Science and Technology, Egypt, Delta University for Science and Technology
Other Study IDs: climate and women health
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-09

CONDITIONS: Women's Health
Keywords: climate change; Women's health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the current study is to assess the impact of climate changes on Women's health.

DETAILED DESCRIPTION:
Climate change is a major global health concern caused by both natural factors and human activities. Climate change including increased exposures to heat, poor air quality, extreme weather events, and altered vector-borne disease transmission, reduced water quality, and decreased food security. These effects directly and indirectly impact human well-being and undermine healthcare services .

Climate change has a significant impact on vulnerable communities, particularly women, who face increased dangers and vulnerabilities. Women often bear the responsibility for managing household affairs and essential resources, but they experience gender disparities in reproductive rights, education, and legal recourse, which are exacerbated during environmental disasters. Sociocultural traditions and familial obligations can prevent women from relocating to safer areas. Additionally, women are disproportionately affected by gender-based violence and are more likely to perish in disasters .

Climate change disproportionally affects women and girls due to systemic gender inequalities. Women's and girls' lower socio-economic status diminishes their ability to cope with climate change. Women represent 70% of the world's poor and are highly dependent on natural resources for their livelihoods. 80% of people displaced by climate change are women.

Women are always seen as caretakers and caregivers in the household settings which makes them vulnerable when they are affected by floods, earthquakes and landslides. There are certain fundamental causes which are affecting women during natural disasters in all aspects as economic, social, ecological, political, physical, and emotional. Extreme weather events disrupt access to essential services by damaging or destroying facilities, infrastructure and medical supply chains, putting many women and girls at greater risk due to having to walk longer distances to access services or not being able to access them at all. o Reduced access to contraception and safe abortion services increases maternal mortality, as well as sexually transmitted infections and unwanted pregnancies.

Egypt aims to create an environment where women and girls can thrive by promoting shared responsibilities, decision-making, and access to sexual and reproductive health services. The National Strategy for the Empowerment of Egyptian Women 2030 outlines key interventions to enhance reproductive health services, raise awareness about risks, and improve healthcare capacities. Climate change was included in the strategy' proposed interventions, to raising women's awareness how to cope and to take necessary protecting procedures, using appropriate environmentally friendly procedures, and training. Egypt's efforts align with the SDGs and demonstrate its commitment to creating a society with equal opportunities and rights for women. A conscious effort needs to be made to raise awareness of these effects and to combat the devastating effects of climate change to our world .Therefore, the current study will be assessing climate change effects on woman's health to disseminating gender-sensitive climate information to communities.

ELIGIBILITY:
Inclusion Criteria:

* Women and girls aging 18 to 60 years
* Working or studying in Al Mansura and Delta university for science and technology and residing in Dakahlia Governorate

Exclusion Criteria:

* known cases of chronic diseases as diabetes mellitus, chronic kidney diseases, hypertension …
* Women diagnosed to have mental illnesses as depression, personality disorders…
* Women residing outside Al Dakahlyea governorate
* Pregnant women

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — women and girls from academic staff, under and postgraduate students, employees and worker's in El Mansoura and delta universities (18-60 years old
Study Population: Sample Size: A representative sample of at least 400 participants will be assigned by simple random sampling technique from academic staff, under and postgraduate students, employees and worker's in El Mansoura and delta universities in the period from 1 august 2024 to the 30 November 2024, sample size was calculated using Open Epi I program at confidence interval 95% and power of 80%.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
increasing awareness of global women climate vulnerability : | 3 months
  1. Sociodemographic and occupational characteristics of women:
     It assesses sociodemographic and occupational characteristics .
  2. women climate vulnerability index: identify 12 risk categories across physical, economic and political sectors that affect women.
  these categories and attendant 51 risk indicators and will require a response on four -point likert rating scale as: one scale for assessing the likelihood of individual risk indicator (Frequent: 0.76-1; Probable: 0.51-0.75; Occasional: 0.26-0.5;Remote: 0-0.25) and one for the impact (Catastrophic: 0.76-1; Signiﬁcant: 0.51-0.75;Moderate: 0.26-0.5; Low: 0-0.25) were used when converting the data into numbers and equations for measuring risk scores.
  Level of risk scores:
  * very high: 7.51-10
  * high :5.01-7.5
  * medium :2.51-5.0
  * low: 0-2.5

SECONDARY OUTCOMES:
increasing Women's health health promoting lifestyle behaviors | 3 months
  health promoting lifestyle behaviors: to measure health promoting lifestyle behaviors (HPLBs). It included fifty-two elements within six dimensions: "Physical activity, nutrition, spiritual growth, interpersonal relations, stress management, and health responsibility". Higher scores refer to higher adherence levels to healthier lifestyle behaviors. The total score ranged from (52 to 208). It used "a four-point likert scale", ranged from one (never) to four (routinely). The total score will be classified into four levels:
  * Poor for the range 52-90
  * Moderate for the range 91-129.
  * Good for the range 130-168.
  * Excellent for the range 169-208.

CONTACTS AND LOCATIONS:
Overall Officials: Basma Wageah elrefay, Lecturer of Nursing, Principal Investigator — Nursing, Faculty of nursing- Delta University for Science and Technology, Egypt
Locations (1):
- Basma Wageah Mohamed Mohamed Elrefay, Mansoura University, Dakahlia Governorate, Egypt

REFERENCES:
- See also: University of Notre Dame. (2021). Rankings // Notre Dame Global Adaptation Initiative // University of Notre Dame. Notre Dame Global Adaptation Initiative. https://gain.nd.edu/our-work/country-index/rankings/ — https://gain.nd.edu/our-work/country-index/rankings/
- See also: Bonnefoi F.(2024) .Sea-Level Rise in the Nile Delta: Promoting Adaptation Through Circular Migration. Baker Institute. https://www.bakerinstitute.org/research/sea-level-rise-nile-delta-promoting-adaptation-through-circular-migration — https://www.bakerinstitute.org/research/sea-level-rise-nile-delta-promoting-adaptation-through-circular-migration